CLINICAL TRIAL: NCT01134328
Title: A Multi-Center, Randomized, Double-Masked Evaluation of the Efficacy of Cetirizine 0.1%/Fluticasone 0.005% Ophthalmic Solution Compared to Its Components and Vehicle in a Modified Conjunctival Allergen Challenge (CAC) Model During Pollen Season
Brief Title: Efficacy of AC-150 for the Treatment of Allergic Conjunctivitis in the Enviro-CAC™ Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aciex Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-100-0005
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- AC-150 Combo (Experimental)
  Interventions: Drug: AC-150 Combo
- AC-150A 0.1% (Active Comparator)
  Interventions: Drug: AC-150A 0.1%
- AC-150B 0.005% (Active Comparator)
  Interventions: Drug: AC-150B 0.005%
- Vehicle (Other)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: AC-150 Combo — 1 drop in each eye for up to 14 days
  Arms: AC-150 Combo
Drug: AC-150A 0.1% — 1 drop in each eye once per day for up to 14 days
  Arms: AC-150A 0.1%
Drug: AC-150B 0.005% — 1 drop in each eye once per day for up to 14 days
  Arms: AC-150B 0.005%
Drug: Vehicle — 1 drop in each eye once per day for up to 14 days
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the efficacy of AC-150 compared to vehicle and its components in the prevention of the signs and symptoms of allergic conjunctivitis in Enviro-CAC™ Model.

ELIGIBILITY:
Inclusion Criteria:

* Positive bilateral conjunctival allergen challenge(CAC) reaction

Exclusion Criteria:

* Known contraindications or sensitivities to the study medication or its components.
* Any ocular condition that, in the opinion of the investigator, could affect the subjects safety or trial parameters.
* Use of disallowed medications during the period indicated prior to study enrollment or during the study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail L Torkildsen, MD, Principal Investigator — Andover Eye Associates; Nicholas P Marsico, MD, Principal Investigator — East West Eye Institute
Locations (1):
- Ora, Inc, Andover, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from two sites in the US.
Pre-assignment Details: There were 83 subjects enrolled, 12 subjects discontinued, and 71 subjects completed the study. Participant flow and baseline characteristics are presented for the 83 subjects that met all inclusion criteria and none of the exclusion criteria and were randomized to receive AC-150 Combo, AC-150A 0.1%, AC-150B 0.005% or Vehicle
Period: Overall Study
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Started | 21 | 21 | 20 | 21
Completed | 19 | 18 | 17 | 17
Not Completed | 2 | 3 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle | Total
Number analyzed (Participants) | 21 | 21 | 20 | 21 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (12.56) | 35.1 (14.32) | 40.2 (12.23) | 38.3 (16.16) | 37.8 (13.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 9 | 10 | 42
  Male | 8 | 11 | 11 | 11 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 3 | 3 | 15
  Not Hispanic or Latino | 17 | 16 | 17 | 18 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 9 | 9 | 7 | 10 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 0 | 0 | 1 | 2
  White | 10 | 9 | 10 | 10 | 39
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 1 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 20 | 21 | 83

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, 7 minutes post-CAC
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 20 | 20 | 19 | 19
units on a scale
  3 minutes post-CAC | 1.33 (0.974) | 0.99 (0.752) | 2.11 (1.173) | 2.90 (0.967)
  5 minutes post-CAC | 1.44 (1.076) | 1.33 (0.590) | 2.25 (1.057) | 3.11 (0.944)
  7 minutes post-CAC | 1.31 (1.033) | 1.59 (0.894) | 2.03 (1.131) | 2.97 (1.018)

2. Primary Outcome: Ocular Itching at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, 7 minutes post-CAC
Population: Intent to Treat (ITT) Population with Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 20 | 19 | 18 | 18
units on a scale
  3 minutes post-CAC | 1.75 (1.112) | 1.92 (1.131) | 1.88 (1.082) | 3.04 (0.693)
  5 minutes post-CAC | 1.95 (1.160) | 2.24 (0.991) | 2.21 (1.132) | 3.18 (0.706)
  7 minutes post-CAC | 1.98 (1.067) | 2.12 (1.156) | 2.11 (1.231) | 3.18 (0.727)

3. Primary Outcome: Ocular Itching at 8 Hours Post-dose at Visit 4A
Description: A treatment efficacy CAC was performed 8 hours after drop instillation. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, 7 minutes post-CAC
Population: Intent to Treat (ITT) Population with Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 20 | 19 | 18 | 18
units on a scale
  3 minutes post-CAC | 1.43 (1.007) | 1.53 (0.916) | 2.01 (0.872) | 2.99 (0.627)
  5 minutes post-CAC | 1.56 (1.022) | 1.83 (0.954) | 2.17 (0.899) | 2.90 (0.703)
  7 minutes post-CAC | 1.64 (1.071) | 1.86 (0.925) | 2.03 (0.935) | 2.79 (0.792)

4. Primary Outcome: Conjunctival Redness at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Conjunctival Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of conjunctival redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT) Population with Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 20 | 19 | 18 | 18
units on a scale
  7 minutes post-CAC | 1.70 (0.677) | 1.97 (0.812) | 2.18 (0.835) | 2.49 (0.639)
  15 minutes post-CAC | 2.04 (0.704) | 2.25 (0.997) | 2.44 (0.770) | 2.58 (0.733)
  20 minutes post-CAC | 2.04 (0.745) | 2.37 (0.980) | 2.51 (0.838) | 2.58 (0.733)

5. Primary Outcome: Conjunctival Redness at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Conjunctival Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of conjunctival redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT) Population with Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 20 | 19 | 18 | 18
units on a scale
  7 minutes post-CAC | 1.56 (0.451) | 1.78 (0.478) | 1.83 (0.485) | 2.01 (0.348)
  15 minutes post-CAC | 1.68 (0.507) | 1.84 (0.410) | 1.97 (0.484) | 2.15 (0.322)
  20 minutes post-CAC | 1.66 (0.424) | 1.88 (0.567) | 1.81 (0.511) | 2.04 (0.386)

6. Primary Outcome: Conjunctival Redness at 8 Hours Post-dose at Visit 4A
Description: A treatment efficacy CAC was performed 8 hours after drop instillation. Conjunctival Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of conjunctival redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Intent to Treat (ITT) Population with Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 20 | 19 | 18 | 18
units on a scale
  7 minutes post-CAC | 1.39 (0.610) | 1.66 (0.560) | 1.81 (0.442) | 1.96 (0.346)
  15 minutes post-CAC | 1.39 (0.626) | 1.70 (0.518) | 1.85 (0.557) | 2.14 (0.366)
  20 minutes post-CAC | 1.44 (0.617) | 1.70 (0.581) | 1.81 (0.546) | 2.14 (0.395)

7. Secondary Outcome: Ciliary Redness at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Ciliary Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ciliary redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 1.44 (0.898) | 1.84 (0.852) | 2.35 (0.834) | 2.37 (0.857)
  15 minutes post-CAC | 1.89 (0.956) | 2.25 (0.940) | 2.47 (0.865) | 2.54 (0.880)
  20 minutes post-CAC | 1.94 (1.100) | 2.29 (0.953) | 2.51 (0.946) | 2.56 (0.788)

8. Secondary Outcome: Ciliary Redness at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Ciliary Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ciliary redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 1.38 (0.577) | 1.81 (0.616) | 1.71 (0.626) | 2.03 (0.499)
  15 minutes post-CAC | 1.51 (0.578) | 1.90 (0.600) | 1.84 (0.712) | 2.10 (0.434)
  20 minutes post-CAC | 1.53 (0.629) | 1.91 (0.637) | 1.72 (0.667) | 2.04 (0.461)

9. Secondary Outcome: Ciliary Redness at 8 Hours Post-dose at Visit 4A
Description: A treatment efficacy CAC was performed 8 hours after drop instillation. Ciliary Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of ciliary redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 1.04 (0.759) | 1.65 (0.673) | 1.68 (0.557) | 2.01 (0.437)
  15 minutes post-CAC | 1.08 (0.702) | 1.69 (0.693) | 1.74 (0.603) | 2.18 (0.393)
  20 minutes post-CAC | 1.15 (0.713) | 1.63 (0.650) | 1.68 (0.717) | 2.10 (0.566)

10. Secondary Outcome: Episcleral Redness at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Episcleral Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of episcleral redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 1.63 (0.749) | 2.03 (0.888) | 2.35 (0.755) | 2.50 (0.667)
  15 minutes post-CAC | 1.90 (0.642) | 2.40 (0.960) | 2.51 (0.763) | 2.71 (0.675)
  20 minutes post-CAC | 1.94 (0.816) | 2.53 (0.951) | 2.56 (0.855) | 2.71 (0.692)

11. Secondary Outcome: Episcleral Redness at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Episcleral Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of Episcleral redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 1.72 (0.575) | 2.12 (0.638) | 2.15 (0.538) | 2.37 (0.516)
  15 minutes post-CAC | 1.79 (0.564) | 2.24 (0.583) | 2.21 (0.663) | 2.53 (0.514)
  20 minutes post-CAC | 1.78 (0.528) | 2.22 (0.522) | 2.16 (0.606) | 2.47 (0.558)

12. Secondary Outcome: Episcleral Redness at 8 Hours Post-dose at Visit 4A
Description: A treatment efficacy CAC was performed 8 hours after drop instillation. Episcleral Redness was assessed by the patient on a 0-4 scale (0=none to 4=severe). Average of episcleral redness score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 1.49 (0.672) | 1.88 (0.644) | 2.04 (0.453) | 2.34 (0.436)
  15 minutes post-CAC | 1.50 (0.712) | 2.04 (0.607) | 2.07 (0.598) | 2.41 (0.484)
  20 minutes post-CAC | 1.57 (0.674) | 1.94 (0.705) | 2.07 (0.630) | 2.40 (0.516)

13. Secondary Outcome: Total Redness at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Total redness was defined as the sum of the conjunctival, ciliary and episcleral redness scores, and was, thus, on a 0-12 scale, making the threshold for clinical significance a treatment difference of 3.0 units. Higher scores represent greater severity.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 4.72 (2.252) | 5.96 (2.450) | 6.99 (2.230) | 7.37 (2.123)
  15 minutes post-CAC | 5.76 (2.225) | 7.03 (2.802) | 7.49 (2.312) | 7.87 (2.208)
  20 minutes post-CAC | 5.86 (2.579) | 7.32 (2.778) | 7.60 (2.631) | 7.88 (2.171)

14. Secondary Outcome: Total Redness at Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Total redness was defined as the sum of the conjunctival, ciliary and episcleral redness scores, and was, thus, on a 0-12 scale, making the threshold for clinical significance a treatment difference of 3.0 units. Higher scores represent greater severity.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 4.60 (1.451) | 5.75 (1.658) | 5.66 (1.591) | 6.40 (1.263)
  15 minutes post-CAC | 4.92 (1.483) | 6.03 (1.489) | 5.88 (1.898) | 6.78 (1.202)
  20 minutes post-CAC | 4.90 (1.402) | 6.10 (1.606) | 5.68 (1.736) | 6.54 (1.312)

15. Secondary Outcome: Total Redness at 8 Hours Post-Dose at Visit 4A
Description: A treatment efficacy CAC was performed 8 hours after drop instillation. Total redness was defined as the sum of the conjunctival, ciliary and episcleral redness scores, and was, thus, on a 0-12 scale, making the threshold for clinical significance a treatment difference of 3.0 units. Higher scores represent greater severity.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 3.83 (1.955) | 5.25 (1.803) | 5.50 (1.389) | 6.29 (1.108)
  15 minutes post-CAC | 3.88 (1.927) | 5.50 (1.730) | 5.63 (1.680) | 6.72 (1.169)
  20 minutes post-CAC | 4.07 (1.905) | 5.35 (1.831) | 5.54 (1.859) | 6.63 (1.415)

16. Secondary Outcome: Lid Swelling at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Lid swelling was assessed by the patient on a 0-3 scale (0=none to 3=severe). Average of lid swelling score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 0.2 (0.43) | 0.5 (0.50) | 1.2 (0.88) | 1.4 (0.63)
  15 minutes post-CAC | 0.4 (0.61) | 0.7 (0.75) | 1.1 (0.97) | 1.5 (0.74)
  20 minutes post-CAC | 0.4 (0.62) | 0.9 (0.75) | 1.1 (0.86) | 1.5 (0.85)

17. Secondary Outcome: Lid Swelling Duration of Action (16 Hours Post-dose)
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Lid swelling was assessed by the patient on a 0-3 scale (0=none to 3=severe). Average of lid swelling score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 0.6 (0.51) | 1.2 (0.95) | 1.1 (0.86) | 1.5 (0.66)
  15 minutes post-CAC | 0.7 (0.59) | 1.3 (1.00) | 1.1 (0.86) | 1.6 (0.70)
  20 minutes post-CAC | 0.7 (0.59) | 1.3 (0.92) | 1.2 (0.95) | 1.7 (0.68)

18. Secondary Outcome: Lid Swelling at 8 Hours Post-dose at Visit 4A
Description: A treatment efficacy CAC was performed 8 hours after drop instillation. Lid swelling was assessed by the patient on a 0-3 scale (0=none to 3=severe). Average of lid swelling score over both eyes was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 0.4 (0.51) | 0.7 (0.58) | 1.1 (1.03) | 1.6 (0.93)
  15 minutes post-CAC | 0.5 (0.50) | 1.0 (0.76) | 1.1 (1.00) | 1.6 (0.70)
  20 minutes post-CAC | 0.5 (0.50) | 1.0 (0.88) | 1.0 (0.94) | 1.6 (0.66)

19. Secondary Outcome: Ear or Palate Pruritus at Onset of Action (15 Minutes Post-dose)
Description: A treatment efficacy CAC was performed 15 minutes after drop instillation. Ear or Palate Pruritus was assessed by the patient on a single 0-4 scale (0=none to 4=severe). Ear or Palate Pruritus score for each time point was analyzed.
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 0.4 (0.78) | 0.3 (0.59) | 0.5 (0.94) | 1.2 (1.39)
  15 minutes post-CAC | 0.4 (0.85) | 0.6 (0.93) | 0.7 (1.10) | 1.4 (1.33)
  20 minutes post-CAC | 0.6 (1.04) | 0.8 (0.90) | 1.0 (1.27) | 1.5 (1.42)

20. Secondary Outcome: Ear or Palate Pruritus at Duration of Action (16 Hours Post-dose)
Description: as for outcome 19
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 0.4 (0.85) | 0.4 (0.62) | 0.4 (0.87) | 1.5 (1.33)
  15 minutes post-CAC | 0.7 (1.13) | 1.3 (0.99) | 0.6 (1.11) | 1.5 (1.37)
  20 minutes post-CAC | 0.7 (1.08) | 1.2 (1.03) | 0.9 (1.43) | 1.5 (1.23)

21. Secondary Outcome: Ear or Palate Pruritus at 8 Hours Post-dose at Visit 4A
Description: as for outcome 19
Time Frame: 7, 15, 20 minutes post-CAC
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 18 | 17 | 17 | 17
units on a scale
  7 minutes post-CAC | 0.3 (0.69) | 0.7 (0.85) | 0.6 (1.06) | 1.2 (1.24)
  15 minutes post-CAC | 0.4 (0.78) | 1.1 (1.05) | 0.8 (1.24) | 1.2 (1.15)
  20 minutes post-CAC | 0.5 (0.86) | 1.2 (1.01) | 0.8 (1.20) | 1.3 (1.16)

22. Secondary Outcome: Tolerability of Study Medication at Visit 2B
Description: Subjects were asked to rate the comfort of the drop in each eye upon instillation, at 1 minute, and at 2 minutes after instillation of study medication. The assessment used a 10-point scale with 0 as very comfortable and 10 as very uncomfortable. Higher scores represent a worse outcome.
Time Frame: upon instillation, 1 minute and 2 minutes post instillation
Population: Intent to Treat (ITT). Number of analyzed subjects differ due to subject discontinuation during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 21 | 21 | 20 | 21
units on a scale
  Upon instillation | 2.3 (1.94) | 2.2 (2.19) | 1.1 (1.54) | 2.0 (1.94)
  1 minute post-instillation | 2.3 (1.59) | 2.0 (2.08) | 0.9 (1.45) | 1.7 (1.55)
  2 minutes post-instillation | 1.9 (1.41) | 1.4 (1.82) | 0.8 (1.25) | 1.6 (1.40)

23. Secondary Outcome: Tolerability of Study Medication at Visit 3
Description: as for outcome 22
Time Frame: upon instillation, 1 minute and 2 minutes post instillation
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Number analyzed (Participants) | 20 | 19 | 18 | 18
units on a scale
  Upon instillation | 2.0 (1.86) | 1.5 (2.12) | 0.9 (1.18) | 1.4 (1.78)
  1 minute post-instillation | 1.6 (1.31) | 1.4 (1.42) | 0.8 (1.06) | 1.0 (1.29)
  2 minutes post-instillation | 1.6 (1.33) | 1.3 (1.25) | 0.7 (0.96) | 0.8 (1.25)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the completion of the study, approximately two months. All subjects who received study medication were evaluable for the safety analysis.
Description: Throughout the visit, staff collected all Adverse Events reported, elicited or observed.
Groups:
- AC-150 Combo: AC-150: 1 drop in each eye for up to 14 days
- AC-150A 0.1%: AC-150A: 1 drop in each eye once per day for up to 14 days
- AC-150B 0.005%: AC-150B: 1 drop in each eye once per day for up to 14 days
Arm/Group | AC-150 Combo | AC-150A 0.1% | AC-150B 0.005% | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes